CLINICAL TRIAL: NCT01344356
Title: Phase IV Trial to Use Stereotactic Body Radiotherapy for Head and Neck Tumors
Brief Title: Stereotactic Body Radiotherapy for Head and Neck Tumors
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mercy Research (Other)
Responsible Party: Principal Investigator, Robert Frazier, MD, Physician, Mercy Research
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-046
Record Dates: First submitted 2011-04-27; First posted 2011-04-29 (Estimated); Results first posted 2020-04-10 (Actual); Last update posted 2020-04-10 (Actual); Status verified 2020-03

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck; Nasopharyngeal Carcinoma; Salivary Gland Cancer; Head and Neck Sarcoma; Paraganglioma of Head and Neck; Chordoma of Head and Neck; Chondrosarcoma of Head and Neck; Angiofibroma of Head and Neck
Keywords: stereotactic radiosurgery; head and neck tumors; squamous cell carcinoma of head and neck
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Nasopharyngeal Carcinoma; Salivary Gland Neoplasms; Head and Neck Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Benign Tumors (Other): Benign head and neck tumors will be treated with SBRT
  Interventions: Radiation: stereotactic body radiotherapy
- Malignant Tumors (Other): Malignant Head and Neck Tumors will be treated with SBRT.
  Interventions: Radiation: Stereotactic body radiotherapy

INTERVENTIONS:
Radiation: stereotactic body radiotherapy — 14-16 Gy / 1 fraction OR 18-21 Gy / 3 fractions (6-7 Gy per fraction)OR 25-45 Gy / 5 fractions (5-9 Gy per fraction)
  Arms: Benign Tumors
Radiation: Stereotactic body radiotherapy — 8-12 Gy / 1 fraction OR 12-18 Gy / 3 fractions (4-6 Gy per fraction) OR 35-45 Gy / 5 fractions (7-9 Gy per fraction)
  Arms: Malignant Tumors

SUMMARY:
This study will evaluate the local control rates as well as acute and late toxicity rates of stereotactic body radiotherapy (SBRT) for the treatment of benign and malignant head and neck tumors.

DETAILED DESCRIPTION:
This single site, non-randomized, prospective, phase IV study includes 3 patient groups to be treated with SBRT:

* Benign tumors, such as paraganglioma, chordoma, chondrosarcoma, as the sole treatment or to gross residual disease after maximal safe resection
* Malignant tumors, such as nasopharynx cancer and squamous cell carcinoma, after initial external beam radiation (Residual Disease Group)
* Unresectable malignant tumors, such as nasopharynx cancer and squamous cell carcinoma, adenocarcinomas, and sarcomas which are recurrent after prior radiation (Primary RT Group) Data collected will include baseline patient demographics, pathology data, radiation therapy procedure, tumor recurrence data, and toxicities.

Follow up data will be collected during the patient's standard office visits. The anticipated duration of this study is 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patient age > 18 years
* Zubrod performance status of 0-3
* Benign head and neck tumors such as paragangliomas, chordoma, chondrosarcoma
* Malignant head and neck cancers such as invasive squamous cell carcinoma, adenocarcinoma, nasopharyngeal carcinoma, salivary gland cancers, and sarcoma
* Signed study-specific consent form

Exclusion Criteria:

* Pregnant or lactating women, due to potential exposure of the fetus to RT and unknown effects of RT on lactating females
* Patients with psychiatric or addictive disorder that would preclude obtaining informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2008-07; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- St. John's Mercy Medical Center, St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Benign Tumors: Benign head and neck tumors will be treated with stereotactic body radiation therapy
  stereotactic body radiotherapy: 14-16 Gray / 1 fraction OR 18-21 Gray / 3 fractions (6-7 Gray per fraction)OR 25-45 Gray / 5 fractions (5-9 Gray per fraction)
- Unrescectable Malignant Tumors: Malignant Head and Neck Tumors will be treated with stereotactic body radiation therapy.
  Stereotactic body radiotherapy: 8-12 Gray / 1 fraction OR 12-18 Gray / 3 fractions (4-6 Gray per fraction) OR 35-45 Gray / 5 fractions (7-9 Gray per fraction)
Period: Overall Study
Arm/Group | Benign Tumors | Unrescectable Malignant Tumors
Started | 1 | 18
Completed | 1 | 9
Not Completed | 0 | 9
Not completed — Physician Decision | 0 | 3
Not completed — Lost to Follow-up | 0 | 6

BASELINE CHARACTERISTICS:
Groups:
- Unrescectable Malignant Tumors: Malignant Head and Neck Tumors will be treated with SBRT.
  Stereotactic body radiotherapy: 8-12 Gy / 1 fraction OR 12-18 Gy / 3 fractions (4-6 Gy per fraction) OR 35-45 Gy / 5 fractions (7-9 Gy per fraction)
- Total: Total of all reporting groups
Arm/Group | Benign Tumors | Unrescectable Malignant Tumors | Total
Number analyzed (Participants) | 1 | 18 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 4 | 4
  >=65 years | 1 | 14 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 0 | 16 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 15 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 3 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1 | 18 | 19

OUTCOME MEASURES:

1. Primary Outcome: Local Control Rate
Description: Complete or partial tumor response or stable disease
Time Frame: 5 years
Population: 12 patients did not have local control rate data reported. 3 patients were enrolled but never treated. 6 patients were lost to follow up. 3 patients died before data was collected.
Measure: Count of Participants; unit: Participants
Arm/Group | Benign Tumors | Malignant Tumors
Number analyzed (Participants) | 1 | 6
Participants | 1 | 5

2. Primary Outcome: Local Recurrence
Description: Instances of progressive disease
Time Frame: 5 years
Population: 12 patients did not have local recurrence rate data reported. 3 patients were enrolled but never treated. 6 patients were lost to follow up. 3 patients died before data was collected.
Measure: Count of Participants; unit: Participants
Arm/Group | Benign Tumors | Malignant Tumors
Number analyzed (Participants) | 1 | 6
Participants | 0 | 3

3. Primary Outcome: Complication Rate
Description: Number of participants with any adverse event
Time Frame: 5 years
Population: 9 patients did not have local control rate data reported. 3 patients were enrolled but never treated. 6 patients were lost to follow up.
Measure: Count of Participants; unit: Participants
Groups:
- Benign Tumors: Benign head and neck tumors will be treated with Stereotactic body radiotherapy
  stereotactic body radiotherapy: 14-16 Gray / 1 fraction OR 18-21 Gray / 3 fractions (6-7 Gray per fraction)OR 25-45 Gray / 5 fractions (5-9 Gray per fraction)
- Unrescectable Malignant Tumors: Malignant Head and Neck Tumors will be treated with Stereotactic body radiotherapy.
  Stereotactic body radiotherapy: 8-12 Gray / 1 fraction OR 12-18 Gray / 3 fractions (4-6 Gray per fraction) OR 35-45 Gray / 5 fractions (7-9 Gray per fraction)
Arm/Group | Benign Tumors | Unrescectable Malignant Tumors
Number analyzed (Participants) | 1 | 9
Participants | 1 | 4

4. Secondary Outcome: Overall Survival
Description: Number of participants who are alive 5 years following treatment.
Time Frame: 5 years
Population: 9 patients did not have overall survival data reported. 3 patients were enrolled but never treated. 6 patients were lost to follow up.
Measure: Count of Participants; unit: Participants
Arm/Group | Benign Tumors | Malignant Tumors
Number analyzed (Participants) | 0 | 10
Participants | 0 | 2

ADVERSE EVENTS:
Time Frame: 5 years
Description: Only events that were considered possibly related to study treatment were recorded as adverse events. Events were graded and categorized using the CTCAE v3.0
Groups:
- Benign Tumors: Benign head and neck tumors will be treated with SBRT
  stereotactic body radiotherapy: 14-16 Gray / 1 fraction OR 18-21 Gray / 3 fractions (6-7 Gray per fraction)OR 25-45 Gray / 5 fractions (5-9 Gray per fraction)
- Malignant Tumors: Malignant Head and Neck Tumors will be treated with SBRT.
  Stereotactic body radiotherapy: 8-12 Gray / 1 fraction OR 12-18 Gray / 3 fractions (4-6 Gray per fraction) OR 35-45 Gray / 5 fractions (7-9 Gray per fraction)
Arm/Group | Benign Tumors | Malignant Tumors
All-Cause Mortality (participants affected / at risk) | 0/1 | 8/10
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/8
Other Adverse Events (participants affected / at risk) | 1/1 | 5/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Benign Tumors (N=1) | Malignant Tumors (N=8)
Esophagitis (Gastrointestinal disorders) | 0 | 2
Mucositis (Gastrointestinal disorders) | 1 | 1
Hoarseness (General disorders) | 0 | 2
Fatigue (General disorders) | 1 | 1
Dizziness (General disorders) | 1 | 0
Cranial Nerve Neuropathy (Nervous system disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2013-02-04): https://cdn.clinicaltrials.gov/large-docs/56/NCT01344356/Prot_000.pdf